CLINICAL TRIAL: NCT05570409
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled TRial Evaluating Immunosuppressive Treatment in Patients With Chronic Virus-Negative Inflammatory cardiomyopaThY (TRINITY Trial)
Brief Title: Immunosuppressive Treatment in Chronic Virus-Negative Inflammatory Cardiomyopathy
Acronym: TRINITY
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Premature end of recruitment due to lack of eligible patients. Within two years of recruitment only nine patients could be randomized out of 130 required patients as per trial protocol.
Sponsor: LMU Klinikum (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); Technical University of Munich (Other); Charite University, Berlin, Germany (Other); University Hospital, Essen (Other); University Hospital Erlangen (Other); University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Steffen Massberg, Prof. Dr. med., LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRINITY
Record Dates: First submitted 2022-09-28; First posted 2022-10-06 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Cardiomyopathy
Keywords: inflammatory cardiomyopathy; heart failure; Mycophenolate mofetil; chronic myocarditis; myocarditis; enomyocardial biopsy; immunosupression
MeSH Terms: conditions — Heart Failure; Myocarditis | interventions — Mycophenolic Acid; Prednisolone

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, multicenter, randomized, double-blind, placebocontrolled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunosuppressive treatment (Experimental): Mycophenolate mofetil (MMF) 1g bid and prednisolone at initially 1mg/kg in a step-down regime
  Interventions: Drug: Mycophenolate Mofetil; Drug: Prednisolone
- Placebo (Placebo Comparator): Mycophenolate mofetil (MMF) and prednisolone Placebo
  Interventions: Drug: Mycophenolate Mofetil Placebo; Drug: Prednisolone Placebo

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Mycophenolate mofetil 1g bid for 6 months
  Other Names: MMF
  Arms: Immunosuppressive treatment
Drug: Prednisolone — initially 1mg/kg in a step-down regime for 6 months
  Arms: Immunosuppressive treatment
Drug: Mycophenolate Mofetil Placebo — MMF matching Placebo
  Other Names: MMF Placebo
  Arms: Placebo
Drug: Prednisolone Placebo — Prednisolone matching placebo
  Arms: Placebo

SUMMARY:
Evaluating Immunosuppressive treatment (Mycophenolate mofetil and prednisolon compared to placebo) for 6 months in patients with chronic virus- Negative Inflammatory cardiomyopathy - a multicenter, randomized, double-blind, placebo-controlled trial.

DETAILED DESCRIPTION:
Inflammatory cardiomyopathy constitutes a relevant part of the cohort of non-dilated left ventricular cardiomyopathy / dilated cardiomyopathy (DCM) and is associated with adverse outcome. Urgent medical needs remain with respect to the therapeutic options for inflammatory cardiomyopathy. So far, no specific therapy for patients with inflammatory cardiomyopathy is available. Existing data on immunosuppression for inflammatory cardiomyopathy is preliminary and needs further validation by larger randomized, controlled, multicenter trials.

Patients with biopsy-proven virus-negative inflammatory dilated or non-dilated left ventricular cardiomyopathy and moderate to severe deterioration of cardiac function despite optimal medical treatment (OMT) for heart failure (HF) will be randomized (1:1) in a double-blinded way to Mycophenolate mofetil (MMF) 1g bid and prednisolone at initially 1mg/kg in a step-down regime for 6 months or placebo. The clinical benefit will be measured with respect to absolute increase in LVEF (metric and binary co-primary endpoints assessed by MRI core lab) of immunosuppressive treatment with MMF and prednisolone compared to placebo at 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Medical therapy for HF for ≥3 months and <10 years according to current guideline recommendations
3. Persistent reduction of LVEF <50% on a routine echocardiographic evaluation (Simpson's biplane) not older than 1 month at time of inclusion
4. EMB with immunohistochemical evidence of lymphocytic myocarditis defined as ≥14 leukocytes/mm2 including up to 4 monocytes/mm2 with the presence of CD3 positive T-lymphocytes ≥7 cells/mm2 and increased MHC-II expression as approved by the histopathology core lab
5. Absence of established cardiotropic virus infection in EMBs (i.e. enteroviruses, HHV-6, EBV, CMV, adenoviruses, parvovirus B19 >500 copies) as approved by the histopathology core lab
6. Negative pregnancy test and the use of a highly effective contraceptive measure in women with child-bearing potential (according to CTFG recommendations)
7. Written informed consent.

Exclusion Criteria:

1. Histopathological (as approved by the histopathology core lab) and/ or clinical evidence of acute lymphocytic myocarditis, sarcoidosis, GCM or eosinophilic myocarditis,
2. Known systemic inflammatory disease,
3. Recent major surgery within <6 weeks, recent ICD implantation within <6 weeks or recent CRT implantation within <3 months prior to,
4. Known coronary artery disease responsible for cardiac dysfunction (i.e., prior myocardial infarction, persistent stenosis ≥ 70%),
5. Pregnancy or lactation,
6. Contraindications to immunosuppressive treatment with MMF + corticosteroids,
7. Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
LVEF increase (metric) | 12 months follow-up
  Absolute increase in LVEF at 12 months follow-up as assessed by blinded investigators of the MRI core lab (metric endpoint)lab) of immunosuppressive treatment with MMF and prednisolone compared to placebo
LVEF increase (binary) | 12 months follow-up
  Proportion of patients with an absolute increase in LVEF ≥10% at 12 months follow-up as assessed by blinded investigators of the MRI core lab (binary endpoint).

SECONDARY OUTCOMES:
Composite clinical outcome | 12 months
  Composite clinical outcome: cardiac death, heart transplantation or a heart failure event (hospitalization for heart failure or the equivalent, i.e., an urgent HF visit) within 12 months from randomization, analyzed as time to first event.physical capacity, cardiac autonomic function, transplant-free survival and hospitalization rate, biomarkers and adverse events
LVEF increase 6 months (MRI) | 6 months follow-up
  Absolute increase in LVEF and rate of increase by ≥10% at 6 months follow-up (MRI, metric, and binary endpoint).
Ventricular remodelling (MRI) | 6 and 12 months follow-up
  Absolute decrease of left ventricular diameters, volumes, mass, and sphericity from baseline to 6 and 12 months follow-up (MRI).
Strain (MRI) | 6 and 12 months follow-up
  Changes in global longitudinal, radial, and circumferential strain from baseline to 6 and 12 months follow-up (MRI).
LVEF increase (echo) | 6 and 12 months follow-up
  Absolute increase in LVEF and rate of increase by ≥10% at 6 and 12 months follow-up (echo, metric, and binary).
Ventricular remodelling (echo) | 6 and 12 months follow-up
  Decrease of left ventricular diameters and volumes by ≥10% at 6 and 12 months follow-up (echo).
Strain (echo) | 6 and 12 months follow-up
  Changes in global longitudinal, radial, circumferential, early, and late diastolic strain (LV), free wall and septal strain (RV), left atrial strain (LA) from baseline to 6 and 12 months follow-up (echo).
Diastolic parameters (echo) | 6 and 12 months follow-up
  Changes in diastolic parameters from baseline to 6 and 12 months follow-up (echo).
Mitral and tricuspid regurgitation (echo) | 6 and 12 months follow-up
  Presence of MR/TR >2 at baseline and at 6 and 12 months followup (echo).
Cardiopulmonary exercise capacity | 6 and 12 months follow-up
  Changes in cardiopulmonary exercise capacity: Distance in the sixminute walk test (6MWT) from baseline to 6 and 12 months followup and (optionally) VO2max, anaerobic threshold and VE/VCO2 on spiroergometry.
NYHA | 6 and 12 months follow-up
  Changes in NYHA functional class from baseline to 6 and 12 months follow-up.
QoL | 12 months
  Changes in patient-reported outcome (quality of life; QOL) from baseline to follow-up as assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ).
Cardiac autonomic function | 6 and 12 months follow-up
  Changes in cardiac autonomic function from baseline to 6 and 12 months follow-up.
Composite safety outcome | 12 months
  Time to the first occurrence of any of the components of the composite safety outcome: death of any cause, arrhythmias requiring intervention, severe adverse events requiring hospitalization.
Biomarker | 12 months
  Time-averaged proportional change in NT-proBNP

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Massberg, Prof Dr. med., Principal Investigator — LMU Klinikum
Locations (14):
- Germany (14):
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Charité - University Hospital Berlin, Berlin
  - University Hospital Essen, Essen
  - UHF- Universitäres Herz- und Gefässzentrum, Frankfurt
  - University Hospital Freiburg - Bad Krozingen, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Göttingen
  - University Hospital Greifswald, Greifswald
  - UKE Hamburg, Hamburg
  - University Hospital Heidelberg, Heidelberg
  - Universitäres Herzzentrum Lübeck, Lübeck
  - Klinikum rechts der Isar, Munich
  - LMU Klinikum, Munich
  - LMU Klinikum Standort Innenstadt, München
  - University Hospital Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: study website — https://trinity.dzhk.de/
- See also: sponsor website — https://www.lmu-klinikum.de/kardiologie/forschung-und-lehre/klinische-forschung/klinische-studien/0890f576db839fe4